CLINICAL TRIAL: NCT01503905
Title: Comparison of the Effectiveness of Neoadjuvant Chemotherapy and the Outcomes Associated With Chemo-induced Amenorrhea Between Docetaxel Plus Epirubicin, and Docetaxel Plus Epirubicin Plus Cyclophosphamide as Neoadjuvant Chemotherapy for Operable Premenopausal Breast Cancer Patients.
Brief Title: Neoadjuvant Chemotherapy for Operable Premenopausal Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Fengxi Su, Director of Department of Breast Tumor Centre, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCSCO001
Record Dates: First submitted 2011-12-29; First posted 2012-01-04 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer Nos Premenopausal
Keywords: breast cancer; neoadjuvant chemotherapy; amenorrhea
MeSH Terms: conditions — Breast Neoplasms; Amenorrhea | interventions — Docetaxel; Epirubicin; Cyclophosphamide; Mastectomy, Modified Radical; Mastectomy, Segmental; Postoperative Period; Radiotherapy; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel plus epirubicin (Active Comparator)
  Interventions: Drug: Docetaxel; Drug: epirubicin; Procedure: Modified radical mastectomy or breast-conserving Surgery; Drug: Docetaxel (post-operative); Drug: Epirubicin (post-operative); Radiation: Radiation therapy; Drug: Herceptin （post-operative); Drug: Tamoxifen (post-operative)
- docetaxel plus epirubicin plus cyclophosphamide (Active Comparator)
  Interventions: Drug: Docetaxel; Drug: epirubicin; Drug: cyclophosphamide; Procedure: Modified radical mastectomy or breast-conserving Surgery; Drug: Docetaxel (post-operative); Drug: Epirubicin (post-operative); Drug: Cyclophosphamide (post-operative); Radiation: Radiation therapy; Drug: Herceptin （post-operative); Drug: Tamoxifen (post-operative)

INTERVENTIONS:
Drug: Docetaxel — 75mg/m2, iv injection, day1, every 21 days
Drug: epirubicin — 80mg/ m2, iv injection, day1, every 21 days
Drug: cyclophosphamide — 500 mg/m2, iv injection, day1, every 21 days
  Arms: docetaxel plus epirubicin plus cyclophosphamide
Procedure: Modified radical mastectomy or breast-conserving Surgery — Two weeks after four cycles of neoadjuvant chemotherapy
Drug: Docetaxel (post-operative) — Two weeks after surgery,75mg/m2, iv injection, day1, every 21 days, 4 cycles totally.
Drug: Epirubicin (post-operative) — Two weeks after surgery, 80mg/m2,iv injection, day1, every 21 days, 4 cycles totally
Drug: Cyclophosphamide (post-operative) — Two weeks after surgery, 500mg/m2, iv injection, day1, every 21 days, 4 cycles totally.
  Arms: docetaxel plus epirubicin plus cyclophosphamide
Radiation: Radiation therapy — Two weeks after post-operative chemotherapy, perform radiation therapy based on 2011 NCCN guideline.
Drug: Herceptin （post-operative) — Perform herceptin therapy (one year) based on 2011 NCCN guideline if the pathological test of the operative tumor sample showed HER2 positive.
Drug: Tamoxifen (post-operative) — After radiation therapy, totally five years. Perform hormone therapy based on 2011 NCCN guideline if the tumor is ER/PR positive.

SUMMARY:
The current study is a multicentre, randomized, open (unblended), prospective clinical trial which is sponsored by the researchers. The trial is designed to compare the effectiveness between docetaxel plus epirubicin, and docetaxel plus epirubicin plus cyclophosphamide as neoadjuvant chemotherapy for operable premenopausal breast cancer patients, and also to compare the outcomes associated with chemo-induced amenorrhea between the two neoadjuvant chemotherapies. The investigators will randomly assign 600 premenopausal female patients with operable breast cancer to receive four cycles of docetaxel and epirubicin (TE); or four cycles of docetaxel, epirubicin, and cyclophosphamide (TEC). After every two cycles of neoadjuvant chemotherapy, the investigators will estimate the effectiveness of therapy. Patients will undergo modified radical mastectomy or breast-conserving surgery after four cycles of neoadjuvant chemotherapy, and then receive postoperative chemotherapy (two cycles), radiation therapy, herceptin targeted therapy or hormone therapy according to the NCCN (2011) guideline. The follow-up will be ten years after surgeries. The primary aim is to examine whether the docetaxel and epirubicin (TE) will be as effective as the docetaxel, epirubicin, and cyclophosphamide (TEC) (pCR rate, cCR rate, PR rate, SD rate, progression-free survival (PFS) and overall survival (OS)). The secondary aim is to correlate chemo (TE/TEC)-induced amenorrhea with outcomes in premenopausal women.

ELIGIBILITY:
Inclusion Criteria:

1. The patients signed the written informed consent.
2. The patients present with operable breast cancers that were diagnosed by histopathology and have no distant metastasis.
3. The patients have no history of anti-cancer therapies including chemotherapy, radiation therapy, hormone therapy and surgical therapy.
4. The patients have normal cardiac functions by echocardiography.
5. The patients' ECOG scores are ≤ 0-2.
6. The age of patient is ≥ 18 years old; And the patients are premenopausal females.
7. The patients are disposed to practice contraception during the whole trial.
8. The results of patients' blood tests are as follows:

   * Hb ≥ 90 g/L
   * WBC ≥ 4.0×109/L
   * Plt ≥ 100×109/L
   * Neutrophils ≥ 1.5×109/L
   * ALT and AST ≤ triple of normal upper limit.
   * TBIL ≤ 1.5 times of normal upper limit.
   * Creatinine ≤ 1.25 times of normal upper limit.

Exclusion Criteria:

1. The patients have other cancers at the same time or have the history of other cancers in recent five years, excluding the controlled skin basal cell carcinoma or skin squamous cell carcinoma or carcinoma in situ of cervix.
2. The patients have active infections that were not suitable for chemotherapy.
3. The patients have severe non-cancerous diseases.
4. The patients are undergoing current administration of anti-cancer therapies, or are attending some other clinical trails.
5. The patients whose breast cancers are HER2 positive and choose to undergo the neoadjuvant chemotherapy that includes herceptin regimen.
6. The patients are pregnant or lactational, or they refuse to practice contraception during the whole trial.
7. The patients are in some special conditions that they can't understand the written informed consent, such as they are demented or hawkish.
8. The patients have allergic history of the chemotherapeutic agents.
9. The patients have bilateral breast cancers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-12; Primary Completion 2018-05 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival of patients. | within 10 years after diagnosis
Overall survival of the patients | within 10 years after diagnosis

SECONDARY OUTCOMES:
The pathological remission rate of patients after neoadjuvant chemotherapy. | within 80 days after diagnosis (after 4 cycles of neoadjuvant chemotherapy)
The clinical remission rate of patients after neoadjuvant chemotherapy | within 80 days after diagnosis (after 4 cycles of neoadjuvant chemotherapy)

CONTACTS AND LOCATIONS:
Overall Officials: Fengxi Su, M.D., Study Chair — Sun Yat-Sen Memerial Hospital of Sun Yat-Sen University
Locations (17):
- China (17):
  - The first People's Hospital of Foshan, Foshan, Guangdong
  - Guangdong Women and Children Hospital, Guangzhou, Guangdong
  - Guangzhou Army General Hospital, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Tumor Hospital of Guangzhou, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Guangzhou Women and Children Hospital, Guangzhou, Guangdong
  - The first People's Hospital of Guangzhou, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Nanfang Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Nanfang Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - The first Affiliated Hospital of Shenzhen University, Shenzhen, Guangdong